CLINICAL TRIAL: NCT05391568
Title: Effects of Dry Needling on Autonomic Nervous System and Nociceptive Pain Processing in Neck Pain. A Randomized Clinical Trial.
Brief Title: Effects of Dry Needling on Autonomic Nervous System and Nociceptive Pain Processing in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015/18
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-05

CONDITIONS: Neck Pain
Keywords: Neck Ache; Cervicalgia; Cervicodynia; Neckache; Cervical Pain; Dry Needling
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Experimental): One single session of DN
  Interventions: Other: Real Dry Needling
- Sham Dry Needling (Sham Comparator): One single session of Sham DN
  Interventions: Other: Sham Dry Needling

INTERVENTIONS:
Other: Real Dry Needling — Needle will be placed at trapezius muscle. "Fast-in, Fast-out" technique will be used at the active trigger point of upper trapezius muscle.
  Arms: Dry Needling
Other: Sham Dry Needling — Sham needle will be placed at trapezius muscle. Simulated "Fast-in, Fast-out" technique will be used at the active trigger point of upper trapezius muscle.
  Arms: Sham Dry Needling

SUMMARY:
Pain in the neck is a musculoskeletal disorder that affects many individuals. Dry needling has shown an effective technique for the treatment of shoulder and neck disorders. The mechanisms of action of the dry needling are not well-known. This study aims to evaluate the effects of dry needling in the upper trapezius on the autonomic nervous system and nociceptive pain processing in patients with non-specific neck pain.

Hypothesis: Dry needling applied in the upper trapezius in patients with non-specific neck pain produced greater activation of the autonomic nervous system and nociceptive pain processing than sham dry needling.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial, using Dry Needling (DN). DN is a technique to treat musculoskeletal pain and physical impairment that consists of introducing needling filaments in the muscle trigger points.

Study Aims:

Aim #1: The primary aim of the study is to compare the effect (during the technique and five minutes after intervention) of a single session of DN on autonomic nervous system as measured by skin conductance in patients with non-specific neck pain with random assignment to two treatments: DN or Sham DN

Aim #2: The secondary aim of the study is to compare the immediate effect on pain sensitivity as measured by pressure pain threshold, activation of descending inhibition pain pathways as measured by temporal summation and conditioned pain modulation in patients with non-specific neck pain with random assignment to two treatments: DN and Sham DN.

Aim #3: The secondary aim of the study is to compare the immediate effect on intensity of pain as numeric pain rating scale (NPRS), relating pain disability (Northwick Park Neck Pain Questionnaire), fear-avoidance of movement (Tampa Scale for Kinesiophobia) and Catastrophizing (Pain Catastrophizing Scale)

Aim #4: The secondary aim of the study is to correlate effects between clinical and other variables.

ELIGIBILITY:
Inclusion Criteria:

1. Pain in the neck area, including the upper trapezius muscle;
2. At least one active TrP (i.e., TrP which referred pain is able to reproduce the patient symptoms in the upper trapezius)
3. Ability to read and understand Spanish
4. Self-reported Intensity of pain rating on the 0-10 NPRS for the neck-shoulder region is 3 or greater
5. Ability to understand, write, and speak Spanish fluently

Exclusion Criteria:

1. Neurological symptoms or signs compatible with cervical radiculopathy or myelopathy
2. Cervical trauma
3. Systemic diseases
4. Pregnancy
5. Psychiatric problems
6. Fear of needles.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Skin Conductance | Through study completion, an average of 20 minutes
  Measured in the hand of the needled upper trapezius. Measured in microsiemens.

SECONDARY OUTCOMES:
Pressure Pain Sensitivity | Baseline; Immediate (10 minutes after intervention)
  Measurement of pressure pain threshold in C5-C6 zygapophyseal joints, dorsal aspect of the midpoint between the base of the nail and the interphalangeal joint of index finger and and the tibialis anterior muscle.
Pressure Pain Stimuli for Temporal Summation | Baseline; Immediate (10 minutes after intervention)
  Measurement of pressure pain stimuli until reach a 6 points in the numeric pain rating scale in the interphalangeal joint of index finger.
Temporal Summation | Baseline; Immediate (10 minutes after intervention)
  Pain response using a numeric pain rating scale will be assessed to pressure stimuli. Series of brief contacts (10 stimuli) of pressure pain threshold will be applied dorsal aspect of the midpoint between the base of the nail and the interphalangeal joint of the index finger.
Conditioned Pain Modulation (CPM) | Baseline; Immediate (10 minutes after intervention)
  CPM will be tested using the lower extremity submaximal effort tourniquet test. Pressure pain threshold (PPT) was assessed using algometry at the dorsal aspect of the midpoint between the base of the nail and the interphalangeal joint at the index finger. After determining the pressure pain threshold (PPT) baseline, the conditioning stimulus was induced using a modified submaximal effort tourniquet procedure.Subjects verbally rated their leg pain until 6 was reached. Although the tourniquet remained inflated, PPT algometry assessment was performed in the same location as previously described (kg/cm2)
Temporal Summation during conditioned stimuli. | Baseline; Immediate (10 minutes after intervention)
  Pain response using a numeric pain rating scale with a 10 scores (0-No pain - 10 The worst pain) will be assessed to pressure stimuli. Series of brief contacts (10 stimuli) of pressure pain threshold will be applied dorsal aspect of the midpoint between the base of the nail and the interphalangeal joint of the index finger using a lower extremity submaximal effort tourniquet test
Pain Intensity (Numeric Pain Rating Scale) | Baseline; one week after intervention
  Pain intensity measured with a 10 scores (0 - No pain - 10 The worst pain) numeric scale
Neck Pain-related Disability | Baseline; one week after intervention
  The Northwick Park Neck Pain (NPQ) assess pain related disability by measuring pain and limitations in the daily activities
Global Rating of Change Scale (GRoC) | One week after intervention
  The patients answered about their perception of improvement during the treatment period on a scale ranging from -7 (a very great deal worse) to zero (about the same) to 7 (a very great deal better).
Kinesiophobia | Baseline; one week after intervention
  The Tampa Scale for Kinesiophobia (TSK-11) was used to evaluate fear of movement and avoidance. Range from 11 to 44 points.
Pain Catastrophizing | Baseline; one week after intervention
  Pain catastrophizing scale (PCS) is a 12-item questionnaire with three components of catastrophizing: magnification, rumination, and helplessness (ranging from 0-52)
Pain Intensity during Intervention (Numeric Pain Rating Scale) | Baseline; immediate (ten minutes after intervention)
  Pain intensity of the intervention was measured on a 10 points numeric pain rating scale (NPRS), 0 (no pain) to 10 (worst pain),

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain